CLINICAL TRIAL: NCT04279210
Title: The Effect of Platelet-rich Plasma on the Female Stress Urinary Incontinence
Brief Title: Platelet-rich Plasma for Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20170048
Record Dates: First submitted 2020-02-16; First posted 2020-02-21 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2017-10

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress urinary incontinence; Platelet-rich plasma
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRP Treatment (Experimental): Women with SUI received PRP injection into anterior vaginal wall (near external urethral sphincter) once per month for three times.
  Interventions: Device: Platelet-rich plasma

INTERVENTIONS:
Device: Platelet-rich plasma — The RegenKit-THT (RegenLab SA, Switzerland) was used to separation of plasma and blood cells. 3mL PRP was extracted from the bottom of the plasma. PRP was injected into anterior vaginal wall, near external urethral sphincter, and into endopelvic fascia.

SUMMARY:
Stress urinary incontinence (SUI) is defined by the International Continence Society (ICS) as "the complaint of any involuntary loss of urine on effort or physical exertion or on sneezing or coughing. The treatment varies from Kegel exercise, bulking agents, vaginal LASER, to surgery. Platelet-rich plasma (PRP) stimulates angiogenesis, promoting vascular in-growth and fibroblast proliferation, enhancing wound-healing in both soft and hard tissue. PRP regulates tissue reconstruction and has been previously used in orthopedics and plastic surgery. The previous study revealed some promising results for PRP use in pelvic floor dysfunction, including SUI. We aim to evaluate the effect of PRP on female SUI.

DETAILED DESCRIPTION:
Women with SUI were enrolled. Pre-treatment evaluation included Overactive Bladder Symptom Score (OABSS), International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI), Pelvic Organ Prolapse Distress Inventory 6 (POPDI-6), Female Sexual Function Index (FSFI), Urinary Distress Inventory Short Form (UDI-6), Incontinence Impact Questionnaire, Short Form (IIQ-7), pelvic examination, and urodynamic study (UDS) (including pad test).

10 milliliter blood was taken from each participant. The RegenKit-THT (RegenLab SA, Switzerland) was used to separation of plasma and blood cells. 3 milliliter PRP was extracted from the bottom of the plasma. PRP was injected into anterior vaginal wall, near external urethral sphincter, and into endopelvic fascia. The participants received one treatment per month for three times. Follow-up schedule is as below: 1st month (transperineal ultrasound and questionnaires), 3rd month (UDS and questionnaires), 6th month (questionnaires), and 12th month (questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* Women with SUI
* Age between 20 to 85 years

Exclusion Criteria:

* Under anti-platelet agent treatment
* Under NSAIDs
* Platelet dysfunction syndrome
* Critical thrombocytopenia
* Hypofibrionogenaemia
* Sepsis
* Acute and chronic infections
* Chronic liver disease
* Anti-coagulation therapy
* History of malignancy
* Pregnancy

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
SUI | 3 months
  The severity of stress urinary incontinence was measured by pad test.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Yu Long, PhD, Principal Investigator — Kaohsiung Municipal University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Result] Billecocq S, Bo K, Dumoulin C, Aigon A, Amarenco G, Bakker E, Cornillet-Bernard M, Cretinon S, Deffieux X, Lartigues G, Loobuick M, Steenstrup B, de Tayrac R. [An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for the conservative and non-pharmacological management of female pelvic floor dysfunction]. Prog Urol. 2019 Mar;29(4):183-208. doi: 10.1016/j.purol.2018.12.010. Epub 2019 Feb 23. French. PMID 30803873
- [Result] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Result] Nygaard I, Barber MD, Burgio KL, Kenton K, Meikle S, Schaffer J, Spino C, Whitehead WE, Wu J, Brody DJ; Pelvic Floor Disorders Network. Prevalence of symptomatic pelvic floor disorders in US women. JAMA. 2008 Sep 17;300(11):1311-6. doi: 10.1001/jama.300.11.1311. PMID 18799443
- [Result] Olsen AL, Smith VJ, Bergstrom JO, Colling JC, Clark AL. Epidemiology of surgically managed pelvic organ prolapse and urinary incontinence. Obstet Gynecol. 1997 Apr;89(4):501-6. doi: 10.1016/S0029-7844(97)00058-6. PMID 9083302
- [Result] Pallua N, Wolter T, Markowicz M. Platelet-rich plasma in burns. Burns. 2010 Feb;36(1):4-8. doi: 10.1016/j.burns.2009.05.002. Epub 2009 Jun 21. PMID 19541423
- [Result] Chrysanthopoulou EL, Pergialiotis V, Perrea D, Kappaourkoulis S, Verikokos C, Doumouchtsis SK. Platelet rich plasma as a minimally invasive approach to uterine prolapse. Med Hypotheses. 2017 Jul;104:97-100. doi: 10.1016/j.mehy.2017.05.018. Epub 2017 May 25. PMID 28673602
- [Result] Shirvan MK, Alamdari DH, Mahboub MD, Ghanadi A, Rahimi HR, Seifalian AM. A novel cell therapy for stress urinary incontinence, short-term outcome. Neurourol Urodyn. 2013 Apr;32(4):377-82. doi: 10.1002/nau.22301. Epub 2012 Sep 12. PMID 22972395
- [Result] Nikolopoulos KI, Pergialiotis V, Perrea D, Doumouchtsis SK. Restoration of the pubourethral ligament with platelet rich plasma for the treatment of stress urinary incontinence. Med Hypotheses. 2016 May;90:29-31. doi: 10.1016/j.mehy.2016.02.019. Epub 2016 Mar 2. PMID 27063081
- [Result] Medel S, Alarab M, Kufaishi H, Drutz H, Shynlova O. Attachment of Primary Vaginal Fibroblasts to Absorbable and Nonabsorbable Implant Materials Coated With Platelet-Rich Plasma: Potential Application in Pelvic Organ Prolapse Surgery. Female Pelvic Med Reconstr Surg. 2015 Jul-Aug;21(4):190-7. doi: 10.1097/SPV.0000000000000178. PMID 25900058